CLINICAL TRIAL: NCT01289210
Title: A Phase I/II Study of Intratumoral Injection of the Small Molecule TLR8 Agonist VTX-2337 in Combination With Local Radiation in Low-Grade B-cell Lymphomas
Brief Title: VTX-2337 in Combination With Radiotherapy in Patients Low-Grade B-cell Lymphomas
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: The study was stopped due to slow rate of recruitment.
Sponsor: Celgene (Industry)
Collaborators: Stanford University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: VRXP-A104; NCT01396018 (obsolete NCT alias)
Record Dates: First submitted 2011-02-01; First posted 2011-02-03 (Estimated); Results first posted 2014-10-06 (Estimated); Last update posted 2019-09-25 (Actual); Status verified 2019-09

CONDITIONS: Low Grade B Cell Lymphoma
Keywords: B cell; lymphoma
MeSH Terms: conditions — Lymphoma | interventions — VTX-2337; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- VTX-2337 plus radiation (Other)
  Interventions: Drug: VTX-2337 plus radiotherapy

INTERVENTIONS:
Drug: VTX-2337 plus radiotherapy — Radiation on Day 1. On Day 2, VTX-2337 3.0mg/m2 is administered intratumorally, followed by radiation. VTX-2337 3.0mg/m2 is then given weekly for 3 weeks in a 4 week cycle over 3 cycles.

SUMMARY:
This study is to determine the safety and effectiveness of VTX-2337 (an investigational drug that stimulates the immune system) in combination with radiation therapy in treating patients with low-grade B-cell lymphoma. Patients will receive 2 low doses of radiotherapy, and 9 intratumoral injections of VTX-2337 over the course of 3 months.

ELIGIBILITY:
Major Inclusion Criteria:

* low grade B cell lymphoma
* 1 or more sites of disease appropriate for intratumoral injection
* measurable disease other than the injection site
* Performance Status of 1 or better
* Adequate bone marrow, renal and hepatic function
* No active autoimmune disease or systemic immunosuppressive drugs
* Life expectancy > 4 months

Exclusion Criteria:

* Known HIV
* Known brain metastases
* Malignancy within last 5 yrs (basal cell or non-invasive squamous cell carcinoma OK)
* Anticoagulation therapy other than 325mg QD ASA
* Significant cardiovascular disease
* Pregnant or nursing

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2011-07; Primary Completion 2011-11 (Actual); Study Completion 2012-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Amar Patel, MD, Study Director — Celgene
Locations (1):
- Stanford Cancer Center, Stanford, California, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- VTX-2337 Plus Radiation: Day 1: radiation therapy; Day 2: VTX-2337 3.0mg/m2 administered intratumorally, followed by radiation. VTX-2337 3.0mg/m2 is then administered weekly for 3 weeks in a 4 week cycle over 3 cycles.
Period: Overall Study
Arm/Group | VTX-2337 Plus Radiation
Started | 2
Completed | 1
Not Completed | 1
Not completed — Adverse Event | 1

BASELINE CHARACTERISTICS:
Arm/Group | VTX-2337 Plus Radiation
Number analyzed (Participants) | 2
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 2
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 2

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Whose Tumors Responded to Treatment With Intratumoral Injection of VTX-2337 in Combination With Low-Dose Local Radiation.
Description: Tumor response was assessed via CT scans of the chest, abdomen, pelvis or other medically appropriate imaging modality to evaluate all areas of disease. Cheson Criteria were used for calculation of response.
Time Frame: Tumor assessment conducted at 12 weeks and every 3-6 months thereafter
Population: Subjects who completed the first 4 weeks of treatment (radiation + 3 VTX-2337 injections) were evaluable for tumor response and immune response. The study was closed due to slow accrual. 2 subjects were enrolled; 1 was evaluable for the primary endpoint, the other discontinued prematurely and was evaluated for safety only (a secondary endpoint).
Measure: Number; unit: participants
Groups:
- VTX-2337 Plus Radiation: Day 1: radiation therapy; Day 2: VTX-2337 3.0mg/m2 administered intratumorally, followed by radiation. VTX-2337 3.0mg/m2 is then admnistered weekly for 3 weeks in a 4 week cycle over 3 cycles.
Arm/Group | VTX-2337 Plus Radiation
Number analyzed (Participants) | 1
participants | 1

2. Secondary Outcome: Assess the Safety and Feasibility of the Combination Regimen.
Time Frame: Safety assessed throughout study period.
Reporting Status: Not Posted

ADVERSE EVENTS:
Arm/Group | VTX-2337 Plus Radiation
Serious Adverse Events (participants affected / at risk) | 0/2
Other Adverse Events (participants affected / at risk) | 2/2
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | VTX-2337 Plus Radiation (N=2)
injection site reaction (General disorders) | 2 (5)
nausea (Gastrointestinal disorders) | 1 (6)
vomiting (Gastrointestinal disorders) | 1 (1)
headache (Nervous system disorders) | 1 (8)
flu like symptoms (General disorders) | 2 (10)
dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
pain (General disorders) | 1 (1)
fatigue (General disorders) | 1/1 (1)
edema - limb (General disorders) | 1 (1)
abdominal pain (Gastrointestinal disorders) | 1 (1)
hypotension (Vascular disorders) | 1 (1)

LIMITATIONS AND CAVEATS:
Due to slow enrollment, the study was closed by the sponsor. 2 participants were enrolled. 1 participant was analyzed for the primary outcome measure (tumor response) and 2 participants were analyzed for safety and toxicity.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No